CLINICAL TRIAL: NCT00216684
Title: An Open Label Study to Confirm the Effectiveness, and Safety of Fentanyl Transdermal Matrix Patch in Japanese Patients With Chronic Intractable Pain Who Has Prior Therapy of Codeine, Morphine Hydrochloride, or Fentanyl Injectable Preparations.
Brief Title: Phase III Clinical Trial of Fentanyl Transdermal Matrix Patch, in the Management of Chronic Intractable Pain- Assessment of Effectiveness, Safety and Pharmacokinetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004879
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Pain, Intractable
Keywords: Fentanyl, Chronic intractable pain, Japanese patients
MeSH Terms: conditions — Pain, Intractable | interventions — Fentanyl

INTERVENTIONS:
Drug: fentanyl

SUMMARY:
The purpose of this study is to verify the effectiveness, and safety in Japanese patients with chronic intractable pain after 4-week medication of fentanyl transdermal matrix patches containing either 12.5 mcg/hr, 25 mcg/hr, 50 mcg/hr, 75 mcg/hr, or 100 mcg/hr, who have been switched from existing formulations, such as codeine, morphine hydrochloride, or fentanyl injectable. Furthermore, the safety and effectiveness of long term treatment such as 48 weeks are to be assessed, if possible.

DETAILED DESCRIPTION:
Fentanyl transdermal matrix patch is a narcotic analgesic agent. Compared with the existing reservoir-type Durotep® Patch, fentanyl transdermal matrix patch is not liable to leakage of drug solution and does not contain alcohol, which becomes a cause of skin irritation. Also this new formulation has become available in a smaller dose of 12.5mg/hr while the smallest Durotep® Patch is 25mg/hr. While Durotep® Patch is currently indicated only for cancer pain in Japan, this clinical trial was planned to assess effectiveness, and safety of fentanyl transdermal matrix patch in Japanese patients with chronic intractable pain receiving codeine, morphine hydrochloride, or fentanyl injectable formulations. After pre-treatment period for seven to fourteen days for evaluating the eligibility of the patients for the study, patients will be treated for 4 weeks as Treatment period 1 and 48 weeks as Treatment period 2 followed by 3-day post-treatment observation period. One patch can be used for 72 hours, which is the same as the existing Patch. Starting from the first day of treatment, fentanyl will be applied to the chest, the upper arm or other appropriate site, which will be replaced with a new patch every three days (ca. 72 hr). Starting dose should be between 12.5 mcg/hr and 75 mcg/hr, depending on the prior opioid dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic intractable pain receiving any of the following treatments :(1)Codeine phosphate, (2)Morphine hydrochloride preparations equivalent to less than 315 mg/day of oral morphine, (3)Fentanyl citrate injectable solution equivalent to less than 0.3 mg/day
* Patients with chronic intractable pain in whom lesions causative of pain cannot be removed or treated, or in whom pain has been persisting for at least 12 weeks despite of the existing medication
* Patients may be hospitalized during application of the initial transdermal dose of fentanyl transdermal matrix patches (patients may be ambulatory when the study starts).

Exclusion Criteria:

* Patients with respiratory dysfunction such as chronic pulmonary disease
* Patients with asthma
* Patients with bradyarrhythmia
* Patients with concurrent liver and/or kidney dysfunction according to the latest laboratory test values within 14 days before the start of the pre-treatment observation period
* Patients with organic brain disorder such as elevated intracranial pressure, disturbance of consciousness/coma, or brain tumor
* Patients with any psychoneurologic complication and judged incapable of self assessment
* Patients with or with a history of drug dependency or narcotic abuse
* Patients with a history of hypersensitivity to fentanyl or any other opioid analgesic

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2005-05; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Patient's global assessments of pain on the completion day of Treatment period 1

SECONDARY OUTCOMES:
Physician's global assessments, pain intensity (Visual Analog Scale: VAS), pain intensity (categorical scale), total pain duration per day, and dose of rescue medication, Adverse events, laboratory values, and vital signs. Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.